CLINICAL TRIAL: NCT00533351
Title: Safety and Efficacy of AGN201781 in Neuropathic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to low enrollment.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 201781-504
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Neuralgia
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AGN201781 (Experimental): AGN201781 50 mg capsules three-time daily for 2 weeks
  Interventions: Drug: AGN201781
- Placebo (Placebo Comparator): placebo 50 mg capsules three-times daily for 2 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AGN201781 — AGN201781 50 mg capsules three-times daily for 2 weeks
  Arms: AGN201781
Drug: placebo — placebo 50 mg capsules three-times daily for 2 weeks
  Arms: Placebo

SUMMARY:
This study will explore the safety and efficacy of AGN201781 in patients with postherpetic neuralgia or post-traumatic peripheral neuralgia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of postherpetic neuralgia or post-traumatic peripheral neuralgia
* Moderate or severe pain associated with postherpetic neuralgia or post-traumatic peripheral neuralgia

Exclusion Criteria:

* Women of child-bearing potential
* Any other uncontrolled diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- St Leonards, New South Wales, Australia
- Kiel, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 2 Treatment Periods in this Cross-Over Study. Patients randomized to AGN201781 during Period 1 received Placebo during Period 2. Patients randomized to Placebo during Period 1 received AGN201781 during Period 2. Period 3 was an Observational Period only (No treatment provided).
Period: Period 1
Arm/Group | AGN201781 Followed by Placebo | Placebo Followed by AGN201781
Started | 7 | 2
Completed | 5 | 1
Not Completed | 2 | 1
Period: Period 2
Arm/Group | AGN201781 Followed by Placebo | Placebo Followed by AGN201781
Started | 5 | 1
Completed | 5 | 1
Not Completed | 0 | 0
Period: Period 3
Arm/Group | AGN201781 Followed by Placebo | Placebo Followed by AGN201781
Started | 3 (Three out of the five patients who completed Period 2 continued to Period 3) | 0 (No patients continued to Period 3)
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN201781 Followed by Placebo | Placebo Followed by AGN201781 | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (11.01) | 49 (36.77) | 54.8 (23.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Subject Global Impression of Change Score at Week 2
Description: Change from baseline in Subject Global Impression of Change score at week 2. The Subject Global Impression of Change is a self-evaluation by the subject of their overall change in relief of neuropathic pain since the beginning of the study rated on a 7-point scale (1=very much improved to 7=very much worse). Due to low number of patients completing the treatment period of the study no analyses were performed.
Time Frame: Baseline, Week 2
Population: Due to low number of patients completing the treatment period of the study no analyses were performed.
Arm/Group | AGN201781 | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change From Baseline in Daily Pain Score at Week 2
Description: Change from baseline in the daily-average-pain score at week 2. This was measured using a 11-point (0 to 10) scale where 0 represented no pain and 10 represented worst pain. Due to the low number of patients completing the treatment period of the study no analyses were performed
Time Frame: Baseline, Week 2
Population: Due to low number of patients completing the treatment period of the study no analyses were performed
Arm/Group | AGN201781 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | AGN201781 Followed by Placebo | Placebo Followed by AGN201781
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 4/7 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN201781 Followed by Placebo (N=7) | Placebo Followed by AGN201781 (N=2)
Fatigue (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1 — Event occurred during Period 3 (Observational/No Treatment)

LIMITATIONS AND CAVEATS:
This study was terminated early due to low enrollment (only 9 of the required 40 subjects had been enrolled). Due to the low number of patients who completed the treatment period of the study, no analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 40 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo